CLINICAL TRIAL: NCT05351957
Title: Dry Needling for Treating Spasticity in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Principal Investigator, Alberto Javier Ormazábal, Physiotherapist, Hospital Universitario de Canarias
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017_100
Record Dates: First submitted 2022-04-21; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis
Keywords: Dry needling, multiple sclerosis, physiotherapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dry Needling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dry needling (Experimental): This study has only 1 arm and the control group is their baseline data
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — Only dry needling of the lower limbs will performed in all patients with acupunture needling

SUMMARY:
The aim of the study is to evaluate the efficacy of dry needling (DN) in the treatment of spasticity in patients with multiple sclerosis (MS). [Participants and Methods] participants with MS, with no evidence of a relapse in the last four weeks and with an EDSS (Expanded Disability Sta- tus Scale) greater than 2.5 points (related with pyramidal score) were recruited. DN was performed in lower limbs for 12 consecutive sessions and evaluated with: EDSS (Pyramidal item), Time up and go (TUG), 25 foot, 9hold peg test (9HPT) and the improvement or not in the quality of life (MSQol54) was verified before and after treatment. A follow up visit was carried out to assess improvement.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient diagnosed with multiple sclerosis.
* Being over 18 years of age and less than or equal to 60 years of age.
* Having a score equal to or greater than 2 in the EDSS.
* They need to have a measurement in the following functional systems: P (pyramidal) >2, CT (brainstem), gait >2 and sphincter >2.
* They need to present hypertonia or contractures of the muscles selected for the dry needling, the pain expressed by the patients must be a consequence of spastic processes, have hourly availability to receive therapies and not have needle phobias.

Exclusion Criteria:

* Having a disease associated with multiple sclerosis that is incompatible with dry needling.
* Being in relapse, or having suffered it in the thirty days prior to starting the treatment. program or taking medications that are contraindicated with the technique applied in the study, (oral anticoagulants.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Change in 9HOLD PEG TEST score | inmediatly before and inmediatly after intervention
  This consists of placing the pegs in the corresponding holes of the 9 holes in the table in the shortest possible time (seconds)
Change in 25 foot walk score | inmediatly before and inmediatly after intervention
  patients must walk a distance of 7.25 meters at the fastest and safest speed for them (seconds)
Change in Time up and go test score | inmediatly before and inmediatly after intervention
  The participants sit in a chair with their backs supported by the back of the chair and their arms resting on the armrests. The participants are asked to get up from the chair and walk a distance of 3 meters, then the patients turn on themselves (360°), walk back to the chair and sit down again (seconds)
Change in Expanded Disability Status Scale (EDSS) score | inmediatly before and inmediatly after intervention
  Each item is valued individually and a score is given, which will then outline the patient's total EDSS ranging from 0 to 10, for use in the exploration sessions. All scans were carried out by a blind explorer.
Change in Multiple sclerosis Quality of life-54 (MSQol54) score | inmediatly before and inmediatly after intervention
  questionnaire of 54 items measuring the quality of life of the patient. It can be self-administered or hetero-administered and both physical and mental aspects are measured. Within these there are subscales: among them quality of life in general. Two summary scores, physical health and mental health, can be derived from a weighted combination of scale scores. They range from 0 to 100, where 100 is the highest quality of life (both for physical and mental health)

CONTACTS AND LOCATIONS:
Overall Officials: MONSERRAT GONZÁLEZ-PLATAS, Study Director — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No